CLINICAL TRIAL: NCT00603239
Title: Safety and Efficacy of Exenatide in Patients With Type 2 Diabetes Using a Thiazolidinedione or a Thiazolidinedione and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWCG
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; metformin; thiazolidinedione; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide twice daily (BID) (Experimental)
  Interventions: Drug: exenatide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5 mcg or 10 mcg, twice a day (BID)
  Other Names: Byetta
  Arms: Exenatide twice daily (BID)
Drug: placebo — subcutaneous injection, volume equivalent to 5 mcg or 10 mcg of active drug, twice a day
  Arms: Placebo

SUMMARY:
This study will assess safety and efficacy of exenatide in combination with a thiazolidinedione (TZD) and a TZD plus metformin over 26 weeks in adult patients with type 2 diabetes who have not achieved adequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* If treated with a thiazolidinedione (TZD) alone, the TZD dose must have been stable for at least 120 days
* The dose of TZD must be: Rosiglitazone (≥4 mg/day) or pioglitazone (≥30 mg/day)
* The metformin dose has been stable for at least 90 days
* Have suboptimal glycemic control as evidenced by an HbA1c between 7.1% and 10.0%, inclusive.
* Have a body mass index (BMI): 25 kg/m2 < BMI < 45 kg/m2.

Exclusion Criteria:

* Have participated in this study previously or any other study using exenatide (AC2993/LY2148568) or glucagon-like peptide-1 (GLP-1) analogs, or have been previously treated with exenatide or GLP-1 analogs
* Have participated in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days of screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.
* Have been treated with exogenous insulin for more than 1 week within the 2 months prior to screening
* Used drugs for weight loss (e.g., orlistat, rimonabant, sibutramine, or similar over-the-counter medications) within 3 months prior to screening.
* Are currently treated with any of the following excluded medications:

  * Sulfonylurea or meglitinide derivatives (e.g., repaglinide or nateglinide) within 3 months prior to screening
  * Alpha-glucosidase inhibitor (e.g., miglitol or acarbose) within 3 months of screening
  * Dipeptidyl peptidase-4 (DPP-4) inhibitors (e.g., sitagliptin or vildagliptin) within 3 months prior to screening
  * Pramlintide acetate injection within 3 months prior to screening
  * Drugs that directly affect gastrointestinal motility, including, but not limited to: Metoclopramide, cisapride, and chronic macrolide antibiotics
  * Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within the 4 weeks immediately preceding study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (25):
- United States (7):
  - Research Site, Birmingham, Alabama
  - Research Site, Concord, California
  - Research Site, Fresno, California
  - Research Site, Denver, Colorado
  - Research Site, Las Vegas, Nevada
  - Research Site, Mogadore, Ohio
  - Research Site, Corvallis, Oregon
- Canada (5):
  - Research Site, New Westminster, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Ajax, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Windsor, Ontario
- Mexico (5):
  - Research Site, Chihuahua City, Chihuahua
  - Research Site, Celaya, Guanajuato
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Mexico City
- Romania (6):
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Dolj
  - Research Site, Iași
  - Research Site, Suceava
- South Africa (2):
  - Research Site, Johannesburg
  - Research Site, Pretoria

REFERENCES:
- [Result] Liutkus J, Rosas Guzman J, Norwood P, Pop L, Northrup J, Cao D, Trautmann M. A placebo-controlled trial of exenatide twice-daily added to thiazolidinediones alone or in combination with metformin. Diabetes Obes Metab. 2010 Dec;12(12):1058-65. doi: 10.1111/j.1463-1326.2010.01251.x. PMID 20977576
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 165 patients, experiencing inadequate glycemic control using a thiazolidinedione (TZD) alone or in combination with metformin, following a 2-week placebo lead-in period, were randomly assigned in a proportion of 2:1 to add exenatide (111 patients) or placebo (54 patients) to their current therapy regimen.
Groups:
- Exenatide Twice Daily (BID): Exenatide 5 mcg twice daily for 4 weeks, followed by 10 mcg twice daily for 22 weeks
- Placebo: Placebo equivalent volume to exenatide 5 mcg for 4 weeks, follwed by placebo equivalent volume to exenatide 10 mcg twice daily for 22 weeks
Period: Overall Study
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Started | 111 | 54
Completed | 96 | 50
Not Completed | 15 | 4
Not completed — Adverse Event | 4 | 1
Not completed — Entry criteria not met | 0 | 1
Not completed — Loss of glucose control | 3 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Subject decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Twice Daily (BID) | Placebo | Total
Number analyzed (Participants) | 111 | 54 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 47 | 144
  >=65 years | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.93 (8.27) | 54.12 (9.36) | 54.67 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 23 | 67
  Male | 67 | 31 | 98

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline to endpoint after 26 weeks of treatment (i.e., HbA1c at endpoint minus HbA1c at baseline)
Time Frame: baseline and 26 weeks
Population: The number of participants was determined based on sample size calculations using parameter estimates from prior study H8O-MC-GWAP (NCT00099320), with change from baseline HbA1c as the primary efficacy measure. Primary analysis is reported for intent to treat population (ITT), last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 110 | 54
Percentage | -0.84 (0.20) | -0.10 (0.23)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline in HbA1c is equal between the two treatment groups. Greater than 99% power to detect a difference between treatment groups of 0.88% in change in HbA1c from baseline using a 2-sided t-test at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustments were made (alpha = 0.05); No adjustments for multiplicity were made

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <= 7%
Description: Percentage of intent-to-treat (ITT) patients who had HbA1c > 7% at baseline that decreased to <= 7% at endpoint (Week 26 or early discontinuation)
Time Frame: 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 104 | 52
percentage of participants | 49.0 | 36.5
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Proportion of subjects with HbA1c <= 7% is equal between the two treatment groups; Test type: Superiority or Other; p = 0.113, CMH test — No adjustments (alpha = 0.05); No adjustment for multiplicity

3. Secondary Outcome: Percentage of Patients Achieving HbA1c <= 6.5%
Description: Percentage of ITT patients who had achieved HbA1c <= 6.5% at endpoint (Week 26 or early discontinuation)
Time Frame: 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 110 | 54
percentage of participants | 33.6 | 13.0
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Proportion of subjects achieving HbA1c <= 6.5% is equal between the two treatment groups; Test type: Superiority or Other; p = 0.004, CMH test — No adjustments (alpha = 0.05); No adjustment for multiplicity

4. Secondary Outcome: Change in Fasting Serum Glucose (FSG)
Description: Change in FSG from baseline to endpoint (26 weeks)
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 103 | 53
mmol/L | -0.65 (0.46) | 0.37 (0.52)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline in FSG is equal between the two treatment groups; Test type: Superiority or Other; p = 0.009, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

5. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to endpoint (26 weeks)
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 111 | 54
kg | -1.43 (0.61) | -0.75 (0.70)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline to endpoint in body weight is equal between the two treatment groups; Test type: Superiority or Other; p = 0.176, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

6. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline to endpoint (26 weeks)
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 109 | 53
cm | -2.26 (3.83) | -1.85 (3.75)

7. Secondary Outcome: Change in Beta-cell Function
Description: Change in homeostatic model assessment-beta cell (HOMA-B) from baseline to endpoint (Week 26) (outcome measure is presented as the ratio of endpoint HOMA-B divided by baseline HOMA-B). HOMA-B is a measure of pancreatic beta-cell function.
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 95 | 49
ratio | 1.08 (0.12) | 0.84 (0.11)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change form baseline in HOMA-B is equal between the two treatment groups; Test type: Superiority or Other; p = 0.009, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

8. Secondary Outcome: Change in Insulin Sensitivity.
Description: Change in homeostatic model assessment-insulin sensitivity (HOMA-S) from baseline to endpoint (26 weeks) (outcome measure is presented as the ratio of endpoint HOMA-S divided by baseline HOMA-S).
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 95 | 49
ratio | 1.09 (0.11) | 1.07 (0.13)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline in HOMA-S is equal between the two treatment groups; Test type: Superiority or Other; p = 0.794, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

9. Secondary Outcome: Number of Subjects Who Experienced an Episode of Minor Hypoglycemia
Description: Overall number of subjects who experienced an episode of minor hypoglycemia.
Time Frame: 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Number; unit: Participants
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 111 | 54
Participants | 4 | 1
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Incidence of minor hypoglycemia episodes is equal between the two treatment groups; Test type: Superiority or Other; p = 1.00, Fisher Exact — No adjustments (alpha = 0.05); No adjustment for multiplicity

10. Secondary Outcome: Change in Impact of Weight on Quality of Life (IWQOL)-Lite Score
Description: IWQOL-Lite analysis of change from baseline to endpoint (26 weeks). IWQOL-Lite is a 31-item questionnaire, assessing the domains of physical function, self-esteem, sexual life, public distress, and work. Response categories for each item range from 1 = "never true" to 5 = "always true."
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 108 | 53
units on a scale
  Change in Total Score | -1.56 (2.21) | 0.11 (2.49)
  Change in Physical Function component | -3.84 (3.06) | -1.05 (3.43)
  Change in Self-Esteem component | 0.20 (2.92) | -0.54 (3.28)
  Change in Sexual Life component | 0.12 (5.52) | 5.01 (6.12)
  Change in Public Distress component | -0.48 (2.61) | -0.28 (2.92)
  Change in Work component | -0.91 (2.41) | 0.08 (2.71)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline in IWQOL-Lite Total Score is equal between the two treatment groups. This statistical analysis is for the Total Score only; Test type: Superiority or Other; p = 0.342, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

11. Secondary Outcome: Change in Euroqol - 5 Domain Quality of Life (EQ-5D) Score
Description: EQ-5D Score - change from baseline to endpoint (26 weeks). EQ-5D is a 5-item questionnaire used to characterize current health states. The tool and accompanying visual analog scale (VAS) assess 5 domains of quality of life, including mobility, self-care, usual activity, pain, and anxiety/depression. Weights are used to score the responses to the 5 domains, with 3 options possible in each domain: extreme problems, some/moderate problems, or no problems. Scores range from 0 to 1, with a score of 1 representing a perfect health state.
Time Frame: baseline and 26 weeks
Population: Based on primary efficacy sample size calculations. Analyses performed on ITT patient population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Number analyzed (Participants) | 108 | 53
units on a scale
  Change in Health State Score | 0.79 (3.54) | -2.94 (3.97)
  Change in Mobility component | 0.14 (0.15) | 0.15 (0.17)
  Change in Self Care component | 0.08 (0.14) | 0.03 (0.16)
  Change Usual Activities component | 0.17 (0.15) | 0.19 (0.17)
  Change in Pain/Discomfort component | 0.29 (0.16) | 0.23 (0.18)
  Change in Anxiety/Depression component | -0.10 (0.16) | -0.26 (0.18)
Statistical Analysis 1: Comparison: Exenatide Twice Daily (BID) vs Placebo; Null hypothesis = Change from baseline in EQ-5D score is equal between the two treatment groups. This statistical analysis is for the EQ-5D Health State Score only; Test type: Superiority or Other; p = 0.186, ANCOVA — No adjustments (alpha = 0.05); No adjustment for multiplicity

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to endpoint, regardless of relationship to study drug. Events were captured as actual terms and coded to MedDRA,version 12.0.
Arm/Group | Exenatide Twice Daily (BID) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/111 | 0/54
Other Adverse Events (participants affected / at risk) | 22/111 | 1/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Twice Daily (BID) (N=111) | Placebo (N=54)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Twice Daily (BID) (N=111) | Placebo (N=54)
Nausea (Gastrointestinal disorders) | 13 | 1
Vomiting (Gastrointestinal disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days